CLINICAL TRIAL: NCT03051100
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Triplet Therapy With Bempedoic Acid (ETC 1002) 180 mg, Ezetimibe 10 mg, and Atorvastatin 20 mg in Patients With Elevated LDL C
Brief Title: Evaluation of the Efficacy and Safety of Bempedoic Acid (ETC-1002) 180mg, Ezetimibe 10mg, and Atorvastatin 20 mg Triplet Therapy in Patients With Elevated LDL-C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1002-038
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Hypercholesterolemia
Keywords: hyperlididemia; LDL; cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Ezetimibe; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Triplet Therapy (Experimental): Bempedoic acid 180 mg, ezetimibe 10 mg, and atorvastatin 20 mg taken orally, daily.
  Interventions: Drug: Bempedoic acid 180mg; Drug: Ezetimibe 10mg; Drug: Atorvastatin 20mg
- placebo (Placebo Comparator): Matching placebos taken orally, daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bempedoic acid 180mg — bempedoic acid 180 mg
  Other Names: ETC-1002
  Arms: Triplet Therapy
Drug: Ezetimibe 10mg — ezetimibe 10 mg
  Other Names: Zetia
  Arms: Triplet Therapy
Drug: Atorvastatin 20mg — atorvastatin 20 mg
  Other Names: Lipitor
  Arms: Triplet Therapy
Other: Placebo — placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if triplet therapy with bempedoic acid (ETC-1002) 180mg, ezetimibe 10mg, and atorvastatin 20mg is effective and safe versus placebo in patients with elevated LDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Fasting LDL-cholesterol between 130 - 189 mg/dL at screening following washout of all LDL-C-lowering drugs and nutritional supplements
* Men and nonpregnant, nonlactating women
* Sufficiently stable and suitable to undergo washout of all LDL-C-lowering drugs and nutritional supplements for 12 weeks

Exclusion Criteria:

* Fasting blood triglycerides greater than or equal to 400 mg/dL
* Body Mass Index (BMI) greater than 50 kg/m2
* History of clinically significant cardiovascular disease
* History of type 1 or type 2 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Haberman, MD, Study Director — Esperion Therapeutics, Inc.
Locations (11):
- United States (11):
  - PMG Research of Christie Clinic, Champaign, Illinois
  - PMG Research of Cary, Cary, North Carolina
  - PMG Research of Charlotte, Charlotte, North Carolina
  - Sensenbrenner Primary Care, Charlotte, North Carolina
  - PMG Research of Hickory, Hickory, North Carolina
  - PMG Research of Raleigh, Raleigh, North Carolina
  - PMG Research of Rocky Mount, Rocky Mount, North Carolina
  - PMG Research Salisbury, Salisbury, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - PMG Research of Charleston, Mt. Pleasant, South Carolina
  - Hampton Roads Center for Clinical Research, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinkosky SL, Newton RS, Day EA, Ford RJ, Lhotak S, Austin RC, Birch CM, Smith BK, Filippov S, Groot PHE, Steinberg GR, Lalwani ND. Liver-specific ATP-citrate lyase inhibition by bempedoic acid decreases LDL-C and attenuates atherosclerosis. Nat Commun. 2016 Nov 28;7:13457. doi: 10.1038/ncomms13457. PMID 27892461
- [Background] Bilen O, Ballantyne CM. Bempedoic Acid (ETC-1002): an Investigational Inhibitor of ATP Citrate Lyase. Curr Atheroscler Rep. 2016 Oct;18(10):61. doi: 10.1007/s11883-016-0611-4. PMID 27663902
- [Background] Thompson PD, MacDougall DE, Newton RS, Margulies JR, Hanselman JC, Orloff DG, McKenney JM, Ballantyne CM. Treatment with ETC-1002 alone and in combination with ezetimibe lowers LDL cholesterol in hypercholesterolemic patients with or without statin intolerance. J Clin Lipidol. 2016 May-Jun;10(3):556-67. doi: 10.1016/j.jacl.2015.12.025. Epub 2016 Jan 6. PMID 27206943
- [Background] Ballantyne CM, McKenney JM, MacDougall DE, Margulies JR, Robinson PL, Hanselman JC, Lalwani ND. Effect of ETC-1002 on Serum Low-Density Lipoprotein Cholesterol in Hypercholesterolemic Patients Receiving Statin Therapy. Am J Cardiol. 2016 Jun 15;117(12):1928-33. doi: 10.1016/j.amjcard.2016.03.043. Epub 2016 Apr 6. PMID 27138185
- [Background] Thompson PD, Rubino J, Janik MJ, MacDougall DE, McBride SJ, Margulies JR, Newton RS. Use of ETC-1002 to treat hypercholesterolemia in patients with statin intolerance. J Clin Lipidol. 2015 May-Jun;9(3):295-304. doi: 10.1016/j.jacl.2015.03.003. Epub 2015 Mar 19. PMID 26073387

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received matching oral placebo once a day.
- Triplet Therapy: Participants received bempedoic acid 180 milligrams (mg), ezetimibe 10 mg, and atorvastatin 20 mg orally once a day.
Period: Overall Study
Arm/Group | Placebo | Triplet Therapy
Started | 20 | 43
Completed | 19 | 43
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Triplet Therapy | Total
Number analyzed (Participants) | 20 | 43 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (7.77) | 61.2 (12.26) | 61.2 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 26 | 40
  Male | 6 | 17 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Black or African American | 3 | 7 | 10
  White | 16 | 34 | 50
Baseline LDL-C, non-HDL-C, HDL-C, TC, and TG Values [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Baseline is defined as the mean of the values from Week -1 (Screening Visit 2) and predose Day 1/Week 0 (Treatment Visit 1). LDL-C, low-density lipoprotein cholesterol. non-HDL-C, non-high-density lipoprotein cholesterol. TC, total cholesterol. TG, triglycerides.
  milligrams per deciliter (mg/dL)
    LDL-C | 155.90 (13.749) | 154.29 (17.913) | 154.80 (16.609)
    non-HDL-C | 183.13 (18.363) | 183.59 (27.347) | 183.44 (24.698)
    HDL-C | 52.03 (12.977) | 52.05 (12.936) | 52.04 (12.844)
    TC | 235.13 (21.196) | 235.67 (26.992) | 235.50 (25.125)
    TG | 139.53 (62.475) | 150.70 (81.375) | 147.15 (75.560)
Baseline Apolipoprotein B (apoB) Values [Mean (Standard Deviation); unit: mg/dL] — Baseline is defined as the predose Day 1/Week 0 (Treatment Visit 1) value.
  mg/dL | 119.2 (15.25) | 118.0 (19.89) | 118.4 (18.42)
Baseline High-Sensitivity C-Reactive Protein (hs-CRP) Values [Median (Full Range); unit: milligrams per Liter] — Baseline is defined as the predose Day 1/Week 0 (Treatment Visit 1) value.
  milligrams per Liter | 1.64 [0.12 to 9.51] | 1.94 [0.27 to 29.16] | 1.88 [0.12 to 29.16]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at Week 6
Description: Percent change from Baseline is calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value ) x 100. Baseline is defined as the mean of the values from Week -1 (Screening Visit 2) and predose Day 1/Week 0 (Treatment Visit 1). Percent change from Baseline in LDL-C was analyzed using analysis of covariance (ANCOVA) with treatment group as a factor and Baseline value as a covariate. Missing LDL-C values were imputed using last observation carried forward (LOCF), with only post-Baseline values carried forward. If LDL-C was measured (i.e., if TG was >400 mg/dL or LDL-C was <50 mg/dL), the measured values were used in the analysis.
Time Frame: Baseline; Week 6
Population: Modified Intent-to-Treat Population: all randomized participants who received at least 1 dose of investigational medicinal product (IMP) and who had a Baseline assessment and at least 1 post-Baseline assessment, excluding any assessment taken more than 2 days after a dose of IMP. Only those participants with data available were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Triplet Therapy
Number analyzed (Participants) | 20 | 43
percent change | -3.1 (3.27) | -63.6 (1.67)
Statistical Analysis 1: Comparison: Placebo vs Triplet Therapy; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -60.5, 95% CI 2-sided [-68.0 to -53.0], Standard Error of Mean 3.67 — Triplet therapy minus placebo

2. Secondary Outcome: Percent Change From Baseline in Lipid Profile Parameters at Week 6
Description: Percent change from Baseline is calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value ) x 100. Baseline is defined as the mean of the values from Week -1 (Screening Visit 2) and predose Day 1/Week 0 (Treatment Visit 1). Baseline apolipoprotein B (apoB) was measured only at predose/Day 1. Percent change from Baseline was analyzed using analysis of covariance (ANCOVA) with treatment group as a factor and Baseline value as a covariate. Missing values were imputed using LOCF, with only post-Baseline values carried forward. non-HDL-C, non-high-density lipoprotein cholesterol; TC, total cholesterol; TG, triglycerides; HDL-C, high-density lipoprotein cholesterol.
Time Frame: Baseline; Week 6
Population: Modified Intent-to-Treat Population. Only those participants with data available were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Triplet Therapy
Number analyzed (Participants) | 20 | 43
percent change
  non-HDL-C: number analyzed (Participants) | 20 | 41
  non-HDL-C | -1.3 (2.56) | -60.0 (1.60)
  TC: number analyzed (Participants) | 20 | 41
  TC | -1.1 (2.24) | -47.1 (1.63)
  apoB: number analyzed (Participants) | 19 | 41
  apoB | 0.6 (2.24) | -53.5 (1.57)
  TG: number analyzed (Participants) | 20 | 41
  TG | 8.9 (5.95) | -27.4 (2.79)
  HDL-C: number analyzed (Participants) | 20 | 41
  HDL-C | 0.4 (2.26) | -1.1 (1.47)
Statistical Analysis 1: Comparison: Placebo vs Triplet Therapy; non-HDL-C; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -58.7, 95% CI 2-sided [-64.9 to -52.6], Standard Error of Mean 3.02 — Triplet therapy minus placebo
Statistical Analysis 2: Comparison: Placebo vs Triplet Therapy; TC; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -46.0, 95% CI 2-sided [-51.6 to -40.4], Standard Error of Mean 2.77 — Triplet therapy minus placebo
Statistical Analysis 3: Comparison: Placebo vs Triplet Therapy; apoB; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -54.1, 95% CI 2-sided [-59.7 to -48.6], Standard Error of Mean 2.74
Statistical Analysis 4: Comparison: Placebo vs Triplet Therapy; TG; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -36.3, 95% CI 2-sided [-49.7 to -22.8], Standard Error of Mean 6.58
Statistical Analysis 5: Comparison: Placebo vs Triplet Therapy; HDL-C; Test type: Superiority; p = 0.588, ANCOVA; Least squares mean difference = -1.5, 95% CI 2-sided [-7.0 to 4.0], Standard Error of Mean 2.7

3. Secondary Outcome: Percent Change From Baseline in High-sensitivity C-reactive Protein (Hs-CRP) at Week 6
Description: Percent change is calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value ) x 100. Baseline is defined as the predose Day 1/Week 0 (Treatment Visit 1) value. If only one value is available either at Week -1 (Screening Visit 2) or Week 0 (Treatment Visit 1), then that value is used as Baseline. Missing values were imputed using LOCF, with only post-Baseline values carried forward.
Time Frame: Baseline; Week 6
Population: Modified Intent-to-Treat Population. Only those participants with data available were analyzed.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Triplet Therapy
Number analyzed (Participants) | 19 | 41
percent change | -2.7 [-19.8 to 17.9] | -47.7 [-66.0 to -22.7]
Statistical Analysis 1: Comparison: Placebo vs Triplet Therapy; Test type: Superiority; p < 0.001, Wilcoxon rank sum test; Median treatment difference = -41.9, 95% CI 2-sided [-60.0 to -21.4], Standard Error of Mean 9.86

4. Secondary Outcome: Number of Participants With LDL-C <70 mg/dL at Week 6
Description: Analysis was based on LOCF values. If LDL-C was measured (i.e., if TG was >400 mg/dL or LDL-C was <50 mg/dL), the measured values were used in the analysis.
Time Frame: Week 6
Population: Modified Intent-to-Treat Population. Only those participants with data available were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Triplet Therapy
Number analyzed (Participants) | 20 | 41
Participants | 0 | 37
Statistical Analysis 1: Comparison: Placebo vs Triplet Therapy; Test type: Superiority; p < 0.001, Fisher Exact

5. Secondary Outcome: Number of Participants With LDL-C Reduction ≥50% From Baseline at Week 6
Description: If LDL-C was measured (i.e., if TG was >400 mg/dL or LDL-C was <50 mg/dL), the measured values were used in the analysis.
Time Frame: Baseline; Week 6
Population: Modified Intent-to-Treat Population. Only those participants with data available were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Triplet Therapy
Number analyzed (Participants) | 20 | 41
Participants | 0 | 39
Statistical Analysis 1: Comparison: Placebo vs Triplet Therapy; Test type: Superiority; p < 0.001, Fisher Exact

ADVERSE EVENTS:
Time Frame: up to 6 weeks plus 30 days
Description: Treatment-emergent adverse events, defined as those events that began or worsened after the first dose of investigational medicinal product (IMP) until 30 days after last dose of IMP, are reported.
Arm/Group | Placebo | Triplet Therapy
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/43
Other Adverse Events (participants affected / at risk) | 7/20 | 15/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | Triplet Therapy (N=43)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 2
Liver function test increased (Investigations) | 0 | 1
Platelet count increased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Principal Investigator plans to publish information from the study, a copy of the manuscript should be provided to the Sponsor for review before submission for publication or presentation. The Sponsor may request that that publication be withheld.

DOCUMENTS (2):
  • Study Protocol (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT03051100/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT03051100/SAP_001.pdf